CLINICAL TRIAL: NCT00059189
Title: Cross-Modal Plasticity of Verbal Memory in the Blind
Brief Title: Brain Plasticity of Verbal Memory in the Blind
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 030163; 03-N-0163
Record Dates: First submitted 2003-04-19; First posted 2003-04-21 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2005-04

CONDITIONS: Blindness
Keywords: Occipital Cortex; Prefrontal Cortex; Transcranial Magnetic Stimulation; Inhibition; Cortical Excitability; Blindness; Healthy Volunteer; HV
MeSH Terms: conditions — Blindness; Inhibition, Psychological

INTERVENTIONS:
Device: Magstim Rapid Magnetic Stimulator

SUMMARY:
This study will examine whether blind people develop changes in the brain that improve memory function. Previous studies have shown that blind people, on average, perform better in memory tasks than sighted people. A possible reason for this is that parts of the brain that process visual information in sighted individuals are engaged in processing mnemonic (remembering) information in blind people.

Blind and sighted people 18 years of age and older are eligible for this study. Healthy, sighted individuals may participate in Part 1 of the study, which is designed to find appropriate words to use in tests for Part 2 of the study. Part 2 will include sighted people and blind people. It will examine whether the (visual) brain in blind people is processing mnemonic information in a way that helps with day-to-day memory functions. Blind participants in this study must have lost their sight by age 4. Candidates will be screened with a medical interview and examination and a brief test of short-term and long-term verbal memory. Sighted patients will also be tested for visual memory and for handedness.

Part 1 - Word Recognition Testing (2 sessions)

* Session 1: Participants listen to a number of words over a loudspeaker and try to remember them for a memory test that will be given 30 minutes later. For the test, subjects listen to words again and press one of three buttons as quickly as possible after hearing the word. The buttons signal whether the subject does or does not recognize the word with a 1) high level of confidence or 2) low level of confidence.
* Session 2: Participants hear a noun over a loudspeaker and have to find an appropriate verb for it, such as the verb (read) for the noun (book).

Part 2 - MRI Scanning and TMS Experiments (5 - 7 sessions)

* Magnetic resonance imaging (MRI): Participants perform the same procedures as described above for Part 1 while undergoing MRI of the brain. For this test, the subject lies on a table inside the MRI scanner - a narrow cylindrical tube with a strong magnetic field. Scanning time varies from 20 minutes to 3 hours, with most scans lasting between 45 and 90 minutes. (Earphones are used to hear the words for this test instead of a loudspeaker.)
* Transcranial magnetic stimulation (TMS): Participants undergo TMS while performing the same procedures described for Part 1. For TMS, a wire coil is held over the scalp. A brief electrical current is passed through the coil, creating a magnetic pulse that stimulates the brain. Subjects may hear a click and feel a pulling sensation on the skin under the coil. There may be a twitch in muscles of the arm or leg. During the TMS, electrical muscle activity is recorded through the electrodes with a computer or other recording device. Each session lasts a maximum of 3 hours.

DETAILED DESCRIPTION:
Cross-modal plasticity refers to the concept that the cortex normally responsive to one sensory modality, when deprived of its usual input, becomes responsive to inputs from other sensory modalities. In blind subjects, the visual cortex processes somatosensory and auditory information. A recent functional imaging study found that verbal memory recall and verb generation significantly activated the primary visual cortex in early blind humans. The magnitude of occipital activation was positively correlated with subsequent performance on verbal memory and verb generation tasks. These results raised the untested hypothesis that the primary visual cortex may be the neural substrate mediating superior verbal memory performance in early blind individuals. The purpose of this protocol is to test this hypothesis.

The first experiment will identify the magnitude of activation in cortical areas associated with successful verbal memory encoding and retrieval, and with verb generation, in blind individuals and sighted controls. The expected outcome is increased involvement of the visual cortex in the early blind group. In the second experiment, we will test the hypothesis that disruption of activity of the activated visual cortex (using TMS) will have deleterious effects on verbal memory encoding and verb generation in early blind subjects, but not in late blind subjects nor sighted controls. The TMS experiment is necessary to identify a cause-effect link between occipital activation and improved memory performance.

Experiment 1: We plan to study early blind subjects, late blind subjects and sighted controls during encoding into and retrieval from episodic verbal memory, and during verb generation, using functional magnetic resonance imaging (fMRI). The primary outcome measure will be the number of voxels significantly activated in primary visual cortex in early blind subjects vs. late blind subjects and sighted controls. Experiment 2: We plan to apply rTMS over left primary visual cortex, left prefrontal cortex, and a control site during encoding of words into and retrieval of words from episodic memory (primary task), and during a verb generation task. Sighted volunteers, early blind and late blind subjects will be studied. The primary outcome measure will be performance on a memory test during rTMS applied to different sites in the different groups. This investigation is important because it can provide novel evidence on a hierarchically high function of the primary visual cortex in the blind.

ELIGIBILITY:
ELIGIBILITY:

Early Blind Subjects: Only compliant early blind subjects who have lost their vision before age 4 years due to diseases affecting the peripheral components of the visual system, i.e., blind subjects without any further neurological problems, and with normal MRI scans, will be selected.

Late Blind Subjects: Only compliant late blind subjects who have lost their vision after age 4 years due to diseases affecting the peripheral components of the visual system, i.e., blind subjects without any further neurological problems, and with normal MRI scans, will be selected.

Sighted Controls: Only compliant adult healthy volunteers with no history of neurological and psychiatric illness who are able to concentrate and to perform simple attentional tasks are eligible.

INCLUSION CRITERIA:

Blind Subjects: Early and late blind subjects (aged 18 or over) will be included in this protocol. Handedness will be assessed by the Edinburgh inventory scale. All experimental sessions will be studied on outpatient basis.

Sighted Subjects: Healthy sighted (normal or corrected-to normal vision) matched in age, sex and level of education to the blind subjects. Handedness will be assessed by the Edinburgh inventory scale.

EXCLUSION CRITERIA:

Exclusion criteria for the study will be any current medical or surgical condition or psychiatric or neurological illness. Furthermore, any individual who is on medication with potential influence on nervous system function, who has a history of surgery with metallic implants or known history of metallic particles in the eye, cardiac pacemaker, intracardiac lines, neural stimulators, cochlear implants, pregnancy, or history of drug abuse, will be excluded from the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 85
Dates: Start 2003-04; Study Completion 2005-04

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Neurological Disorders and Stroke (NINDS), Bethesda, Maryland, United States

REFERENCES:
- [Background] Alho K, Kujala T, Paavilainen P, Summala H, Naatanen R. Auditory processing in visual brain areas of the early blind: evidence from event-related potentials. Electroencephalogr Clin Neurophysiol. 1993 Jun;86(6):418-27. doi: 10.1016/0013-4694(93)90137-k. PMID 7686476
- [Background] Bridgers SL, Delaney RC. Transcranial magnetic stimulation: an assessment of cognitive and other cerebral effects. Neurology. 1989 Mar;39(3):417-9. doi: 10.1212/wnl.39.3.417. PMID 2927652
- [Background] Burton H, Snyder AZ, Diamond JB, Raichle ME. Adaptive changes in early and late blind: a FMRI study of verb generation to heard nouns. J Neurophysiol. 2002 Dec;88(6):3359-71. doi: 10.1152/jn.00129.2002. PMID 12466452